CLINICAL TRIAL: NCT01626664
Title: Multi-Center, Open-Label, Randomized Study of Anti-CCR4 Monoclonal Antibody KW-0761 or Investigator's Choice in Subjects With Previously Treated Adult T-cell Leukemia-Lymphoma (ATL)
Brief Title: KW-0761 or Investigator's Choice in Subjects With Previously Treated Adult T-cell Leukemia-Lymphoma (ATL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROTOCOL 0761-009
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Adult T-cell Leukemia-Lymphoma
Keywords: Adult T cell Leukemia-Lymphoma (ATL)
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — mogamulizumab; 10-propargyl-10-deazaaminopterin; Gemcitabine; Oxaliplatin; Calcium Dobesilate; Dexamethasone; Cisplatin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KW-0761 (Experimental): anti-CCR4 monoclonal antibody KW-0761 (mogamulizumab)
  Interventions: Biological: KW-0761
- investigator's choice (Active Comparator): Comparator is investigator's choice of pralatrexate or gemcitabine plus oxaliplatin or DHAP
  Interventions: Drug: Pralatrexate; Drug: gemcitabine plus oxaliplatin; Drug: DHAP

INTERVENTIONS:
Biological: KW-0761 — 1.0 mg/kg weekly x 4 in cycle 1 then every other week until progression
  Other Names: mogamulizumab; POTELIGEO®
  Arms: KW-0761
Drug: Pralatrexate — 30 mg/m2 weekly for 3 weeks followed by 1 week of no therapy until progression
  Other Names: Folotyn
  Arms: investigator's choice
Drug: gemcitabine plus oxaliplatin — gemcitabine 1000 mg/m2, followed by oxaliplatin 100 mg/m2 every 2 weeks until progression
  Other Names: Gemzar; Eloxatin; GemOx
  Arms: investigator's choice
Drug: DHAP — dexamethasone 40 mg on Day 1-4, cisplatin 100 mg/m2 on Day 1 followed by 2 doses of cytarabine 2000 mg/m2 every 4 weeks until progression
  Other Names: Decadron, Dexasone, Baycadron; Platinol; Depocyt, Ara-C
  Arms: investigator's choice

SUMMARY:
The purpose of this study is to estimate the overall response rate of subjects with relapsed or refractory Adult T-cell Leukemia-Lymphoma (ATL).

DETAILED DESCRIPTION:
CCR4 expression in ATL patients has been demonstrated to be very high and has been associated with shorter survival compared with CCR4-negative patients. KW-0761, a monoclonal antibody targeted to CCR4, has been shown to be safe and tolerable in several clinical trials in subjects with a variety of T-cell malignancies, including ATL, mycosis fungoides and Sézary syndrome. The objective of this study is to estimate the overall response rate of KW-0761 for subjects with relapsed or refractory ATL.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects ≥ 18 years of age
* Confirmed diagnosis of ATL (excluding smoldering subtype)
* Subjects must currently have evidence of disease in at least one of the following:

  * Lymph nodes
  * Extranodal masses
  * Spleen or liver
  * Skin
  * Peripheral blood
  * Bone marrow
* Relapsed or refractory after at least one prior systemic therapy regimen for ATL;
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2 at study entry
* Resolution of all clinically significant toxic effects of prior cancer therapy to grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI-CTCAE, v.4.0)
* Adequate hematological, hepatic and renal function

Exclusion Criteria:

* Smoldering subtype of ATL;
* Lymphomatous or acute subtype subject with > 2 prior systemic therapy regimens and who has not achieved a response (CR or PR) or maintained stable disease for at least 12 weeks on last immediate prior therapy;
* History of allogeneic transplant;
* Autologous hematopoietic stem cell transplant within 90 days of study entry;
* Untreated human immunodeficiency virus (HIV)
* Has known hepatitis C. Patients who are hepatitis C antibody positive but are hepatitis C quantitative PCR negative may be enrolled;
* Has hepatitis B based on PCR testing for hepatitis B virus DNA. Patients who are hepatitis B core antibody positive but PCR negative may be enrolled if placed on appropriate anti-hepatitis B virus prophylaxis prior to commencing treatment with KW-0761. Patients who are hepatitis B core antibody positive based on prior vaccination need not receive prophylaxis;
* Have had a malignancy in the past two years except non-melanoma skin cancers, melanoma in situ, localized cancer of the prostate with current PSA < 0.1 µg/mL, treated thyroid cancer or cervical carcinoma in situ or ductal/lobular carcinoma in situ of the breast who is currently without evidence of disease;
* Clinical evidence of central nervous system (CNS) involvement or metastasis. In subjects suspected of having CNS disease, an MRI of the brain and/or lumbar puncture should be done to confirm;
* Psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit compliance with study requirements;
* Significant uncontrolled intercurrent illness
* Experienced allergic reactions to monoclonal antibodies or other therapeutic proteins;
* Known active autoimmune diseases will be excluded (For example; Grave's disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease);
* Is pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or lactating.
* Prior treatment with KW-0761;
* Initiation of treatment with systemic corticosteroids while on study is only permitted for acute and brief complications of underlying disease (e.g., hypercalcemia) or for treatment related side effects (e.g., including pre-medication for infusion reaction, nausea and vomiting). Subjects on systemic corticosteroids prior to enrollment must be off for 7 days before initiation of study treatment, unless specifically indicated for the treatment of hypercalcemia. (subjects may receive inhalation corticosteroids and replacement doses of systemic corticosteroids as needed);
* Initiation of treatment with topical corticosteroids while on study is not permitted except to treat an acute rash. Subjects on a stable dose of medium or low potency topical corticosteroids for at least 4 weeks prior to Pre-treatment Visit may continue use at the same dose, although the investigator should attempt to taper the use to lowest dose tolerable;
* Have had interferon-α and/or zidovudine within 1 week, or anti-neoplastic chemotherapy, radiation, immunotherapy, or investigational medications within 2 weeks of first study treatment;
* Subjects on any immunomodulatory drug. Subjects on any immunomodulatory drug within 4 weeks of their first dose of KW-0761 are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (20):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Miami / Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering, New York, New York
  - Columbia Presbyterian, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Brazil (2):
  - Hospital Universitario Professor Edgard Santos- UFBA, Salvador, Bahia
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Sao Paulo- SP
- France (2):
  - CHU de Fort de France, Fort de France Cedex
  - Hospital Necker, Paris
- Peru (2):
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Instituto Oncologico Miraflores, Lima
- United Kingdom (3):
  - Guy's Hospital, London
  - Imperial College, London
  - Sandwell General Hospital, West Midlands

RESULTS

PARTICIPANT FLOW:
Groups:
- IC Original Then Crossover to KW-0761: Subjects who were randomized to the Investigator's Choice regimen could be crossed over to receive mogamulizumab upon disease progression and with permission from the Medical Monitor.
Period: Randomization Period
Arm/Group | KW-0761 | Investigator's Choice | IC Original Then Crossover to KW-0761
Started | 47 | 24 | 0
Completed | 47 | 24 | 0
Not Completed | 0 | 0 | 0
Period: Crossover Period
Arm/Group | KW-0761 | Investigator's Choice | IC Original Then Crossover to KW-0761
Started | 0 | 0 | 18
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KW-0761 | Investigator's Choice | Total
Number analyzed (Participants) | 47 | 24 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 22 | 57
  >=65 years | 12 | 2 | 14
Age, Continuous [Mean (Full Range); unit: years] | 55 [22 to 82] | 49 [24 to 80] | 53 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 24 | 10 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 31 | 14 | 45
  Unknown or Not Reported | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6 | 5 | 11
  Race: Asian | 2 | 1 | 3
  Race: Black or African American | 32 | 15 | 47
  Race: Other | 1 | 0 | 1
  Race: Not Applicable | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 25 | 14 | 39
  Brazil | 3 | 0 | 3
  United Kingdom | 9 | 4 | 13
  France | 6 | 3 | 9
  Peru | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate was determined based on the response in all compartments (lymph nodes, extranodal masses, spleen/liver, skin, peripheral blood, and bone marrow), referencing Tsukasaki, 2009 as follows: Complete Response (CR) = All compartments involved with disease must be CR; Uncertified Complete Response (CRu) = > 75% decrease in lymph nodes and/or extranodal disease with all other compartments involved with disease CR; Partial Response (PR) = If any compartment is CR/PR and all other compartments involved with disease are at least SD; Stable Disease (SD) = All compartments involved with disease are SD; Progressive Disease (PD) = PD in any compartment.
  Lymph node and extranodal masses response ≥50% decrease by CT, skin response ≥50% decrease in mSWAT score; blood response ≥50% decrease in malignant cells by flow cytometry; normal bone marrow if abnormal at baseline. PD equals New or ≥50% increase in any compartment.
Time Frame: every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first
Measure: Number; unit: participants
Arm/Group | KW-0761 | Investigator's Choice
Number analyzed (Participants) | 47 | 24
participants
  Complete Response | 2 | 0
  Uncertified Complete Response | 0 | 0
  Partial Response | 11 | 2
  Stable Disease | 0 | 4
  Relapsed Disease or Progressive Disease | 16 | 13
  Not Assessable | 18 | 5
  Overall Response Rate (Confirmed and Unconfirmed) | 13 | 2
  Overall Response Rate Confirmed | 5 | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival was defined as the time from the first date of treatment until the date that PD or death was first reported. Disease progression included PD in any compartment per ATL response criteria, clinical progression at the end of the randomized treatment, or disease progression reported during the follow-up period. The date of PD was the earliest date at which disease progression could be declared.
Time Frame: From date of randomization until the date of first documented progression, start of alternative therapy, or date of death from any cause, whichever came first, up to 36 months
Measure: Median (95% Confidence Interval); unit: percentage of subjects
Arm/Group | KW-0761 | Investigator's Choice
Number analyzed (Participants) | 47 | 24
percentage of subjects
  PFS Subjects (%) Alive for at Least: 1 Month | 47.5 [31.6 to 61.9] | 44.1 [22.8 to 63.4]
  PFS Subjects (%) Alive for at Least: 2 Months | 29.8 [16.6 to 44.2] | 33.0 [14.2 to 53.3]
  PFS Subjects (%) Alive for at Least: 3 Months | 24.4 [12.4 to 38.5] | 26.4 [9.4 to 47.3]
  PFS Subjects (%) Alive for at Least: 4 Months | 18.3 [7.9 to 32.1] | 13.2 [2.4 to 33.5]
  PFS Subjects (%) Alive for at Least: 5 Months | 18.3 [7.9 to 32.1] | 0 [0 to 0]
  PFS Subjects (%) Alive for at Least: 6 Months | 12.2 [4.0 to 25.1] | 0 [0 to 0]

3. Secondary Outcome: Overall Survival
Description: The estimates and summary statistics for OS were calculated based on Kaplan-Meier method, and the median OS was 4.9 months for subjects randomized to the mogamulizumab group versus 6.87 months for subjects randomized to the Investigator's Choice group.
Time Frame: up to 36 months
Measure: Median (95% Confidence Interval); unit: percentage of subjects
Arm/Group | KW-0761 | Investigator's Choice
Number analyzed (Participants) | 47 | 24
percentage of subjects
  Subjects (%) Alive for at Least: 1 Month | 87.0 [73.2 to 93.9] | 91.7 [70.6 to 97.8]
  Subjects (%) Alive for at Least: 2 Months | 75.6 [60.3 to 85.7] | 79.2 [57.0 to 90.8]
  Subjects (%) Alive for at Least: 3 Months | 59.1 [43.1 to 72.0] | 70.8 [48.4 to 84.9]
  Subjects (%) Alive for at Least: 4 Months | 54.3 [38.5 to 67.7] | 66.7 [44.3 to 81.7]
  Subjects (%) Alive for at Least: 5 Months | 49.5 [33.9 to 63.3] | 54.2 [32.7 to 71.4]
  Subjects (%) Alive for at Least: 6 Months | 44.3 [29.1 to 58.5] | 54.2 [32.7 to 71.4]

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Total Score
Description: The FACT-Lym consists of a 27-item general core questionnaire (i.e., Functional Assessment of Cancer Therapy - General [FACT-G]) and a 15-item disease-specific questionnaire (Lymphoma Subscale). The FACT-G includes 4 domains: physical well-being, social/family well-being, emotional well-being, and functional well-being. The total FACT-Lym score (0-168) was obtained by summing individual subscale scores. Higher scores for the scales indicate better quality of life. Change was calculated as the value at the last observation minus the value at baseline.
Time Frame: From date of randomization until the date of first documented progression, up to 36 months
Population: All participants in Intention-to-Treat who had both the values at baseline and last observation
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KW-0761 | Investigator's Choice
Number analyzed (Participants) | 41 | 24
Units on a scale
  Baseline: number analyzed (Participants) | 41 | 21
  Baseline | 110.1 (22.15) | 106.8 (25.84)
  Last Observation Change from Baseline: number analyzed (Participants) | 27 | 14
  Last Observation Change from Baseline | -12.1 (25.60) | -14.9 (25.56)

ADVERSE EVENTS:
Time Frame: From pre-treatment visit until 90 days after the last dose, approximately three months overall
Arm/Group | KW-0761 | Investigator's Choice | IC Original Then Crossover to KW-0761
All-Cause Mortality (participants affected / at risk) | 10/47 | 1/24 | 12/18
Serious Adverse Events (participants affected / at risk) | 26/47 | 10/24 | 9/18
Other Adverse Events (participants affected / at risk) | 45/47 | 24/24 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=47) | Investigator's Choice (N=24) | IC Original Then Crossover to KW-0761 (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemsis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Multi-Organ Failure (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective Thrombosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Post Procedural Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Amylase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine Ketone Body Present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Osmotic Demyelination Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Plerual Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=47) | Investigator's Choice (N=24) | IC Original Then Crossover to KW-0761 (N=18)
Anaemia (Blood and lymphatic system disorders) | 10 (13) | 3 (10) | 6 (11)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (10) | 4 (8) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8) | 3 (5) | 2 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (7) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (9) | 2 (2)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 9 (11) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6) | 7 (7) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (8) | 4 (4) | 1 (1)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 8 (8) | 4 (4) | 3 (3)
Pain (General disorders) | 3 (3) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 6 (18) | 3 (3)
Aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 21 (23) | 0 (0) | 8 (8)
Alanine Aminotransferase Increased (Investigations) | 3 (4) | 2 (12) | 0 (0)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Aspartate Aminotransferase Increased (Investigations) | 5 (5) | 2 (13) | 2 (2)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 3 (8) | 1 (1)
Blood Bicarbonate Decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood Creatinine Increased (Investigations) | 5 (5) | 2 (2) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 6 (7) | 1 (1) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Neutrophil Count Decreased (Investigations) | 2 (3) | 4 (4) | 1 (2)
Platelet Count Decreased (Investigations) | 5 (5) | 2 (11) | 0 (0)
Platelet Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Urine Output Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (8) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (8) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (5) | 2 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (5) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (7) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (5) | 3 (10) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 3 (3) | 1 (2)
Headache (Nervous system disorders) | 4 (4) | 7 (7) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Confusional State (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Renail Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Sexual Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 9 (15) | 0 (0) | 4 (6)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less